CLINICAL TRIAL: NCT05605938
Title: Multicenter Double-blind Placebo-controlled Randomized Clinical Trial of the Efficacy and Safety of Tenoten for Children in 12-week Treatment of Children With Anxiety Disorders
Brief Title: Efficacy and Safety of Tenoten in the Treatment of Children With Anxiety Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-TD-001
Record Dates: First submitted 2022-10-25; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-05

CONDITIONS: Anxiety Disorder of Childhood
MeSH Terms: interventions — tenoten

STUDY DESIGN:
Intervention Model Description: double-blind placebo-controlled randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenoten for children (Experimental): 1 tablet 3 times daily for 12 weeks. Route of administration: sublingual, the tablet should be held in the mouth until completely dissolved.
  Interventions: Drug: Tenoten for children
- Placebo (Placebo Comparator): As per the Tenoten for children dosing regimen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tenoten for children — Oral administration
  Arms: Tenoten for children
Drug: Placebo — Oral administration
  Arms: Placebo

SUMMARY:
Purpose of the study:

• evaluate the efficacy and safety of Tenoten for children in children with anxiety disorders.

DETAILED DESCRIPTION:
Design: a multicenter, double-blind, placebo-controlled, parallel-group randomized clinical trial.

The study includs children of both sexes aged 5 to 15 years who were diagnosed by a neurologist with an anxiety disorder (according to the ICD-10, one of the variants of an emotional disorder with an onset specific to childhood - F 93).

After a parent/legal representative signed an informed consent form for participation in the clinical trial at the screening visit (Visit 1, Day 0), patients underwent an initial examination, including medical history, assessment of vital signs, and physical examination; concomitant therapy was recorded. The initial severity of anxiety disorders (from mild to severe) was assessed using a scale for assessing the severity of anxiety in children (G.P. Lavrentieva, T.M. Titarenko), using an anxiety test (R. Temple, V. Amen, M. Dorki) and Spence Children's Anxiety Scale (SCAS). If the inclusion criteria were met and no exclusion criteria were met, the patient was included in the study and randomized to one of the groups: Tenoten for children or Placebo (day 0, visit 1). In the course of treatment, patients made 3 visits to the doctor within 12 weeks (at 4, 8 and 12 weeks), during which the dynamics of the severity of anxiety disorders were recorded using an anxiety test (R. Temple, V. Amen, M. Dorki) and SCAS; vital signs and physical examination were performed, prescribed and concomitant therapy were controlled. At visit 4 (week 12), doctor assessed the therapeutic dynamics and treatment side effects by the end of the treatment period in scores on the Clinical Global Impression (CGI) scale.

ELIGIBILITY:
Inclusion Criteria:

1. Children of both sexes aged 5 to 15 years inclusive.
2. At least one of the diagnoses from ICD-10 Diagnosis Code F 93 - Emotional disorders with onset specific to childhood:

   * Separation anxiety disorder of childhood - F 93.0;
   * Phobic anxiety disorder of childhood - F 93.1;
   * Social anxiety disorder of childhood - F 93.2;
   * Generalized anxiety disorder of childhood - F 93.8.
3. Mild to severe disease, with the severity assessed using the following scales:

   * Child Anxiety Scale of G.P. Lavrentieva and T.M. Titarenko;
   * anxiety test of R. Temple, V. Amen, M. Dorky;
4. No signs of severe cognitive development deficiency, according to the investigator;
5. No drug treatment for anxiety disorders within the last two weeks;
6. Availability of singed informed consent from the legal representative of a child. In addition, patients aged ≥14 years are to sign a patient informed consent form.

Exclusion Criteria:

1. Age under 5 or over 15 years;
2. Decompensated somatic diseases that may affect the conduct of the trial;
3. Severe residual signs of organic CNS injury;
4. Hallucinations, delusions, and psychotic affective disorders;
5. Mental retardation and oligophrenic-like impairment;
6. Hypersensitivity to any components of the study drugs;
7. Reluctance of a child or his/her legal representatives to participate in the clinical study;
8. The patient's legal representative with drug abuse problems, alcoholism, or mental disorders;
9. Participation in other clinical studies within 4 months prior to enrollment in the current trial.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2010-07-28 (Actual); Primary Completion 2011-10-28 (Actual); Study Completion 2011-10-28 (Actual)

PRIMARY OUTCOMES:
Changes in SCAS scores | 12 weeks
  Spence Children's Anxiety Scale (SCAS).The study uses 3 scales: (1) for patients aged 5-7 years and (2) for patients aged 8-15 (both of them filled in by patient's legal representatives); (3) for patients aged 8-15 years (filled in by patient).
  Maximum total score of each scales is 114. A higher score reflects a higher level of anxiety
Changes in severity of anxiety according to test of R.Temple, V.Amen, M.Dorky | 12 weeks
  The questionnaire is filled in by legal representative of patient. Each "yes" answer means 1 point. Severe anxiety 15-20 points; moderate 7-14 points; mild 1-6 points
Percentage of patients who progress to milder anxiety disorders | 12 weeks
  Based on medical records

SECONDARY OUTCOMES:
Changes in anxiety disorder symptoms according to SCAS domains, depending on type of anxiety disorders | 12 weeks
  Based on medical records
Comparison of mean CGI scores between study groups | 12 weeks
  Clinical Global Impression (CGI) scale consists of three subscales: severity of condition, overall degree of its improvement on 7-point system, and subscale of the efficacy index, which is calculated from the combination of one of four degrees of therapeutic effect (noticeable, moderate, minimal, no change) and severity of the side effect drug (absent, insignificant, significant, leveling therapeutic effect)
Occurrence and characteristics of adverse events | 12 weeks
  Based on medical records. Occurrence, severity, relationship with medicine, outcomes of adverse events

CONTACTS AND LOCATIONS:
Locations (5):
- Russia (5):
  - Specialized Clinical Psychiatric Hospital # 1, Krasnodar
  - Scientific Center for Mental Health of the Russian Academy of Medical Sciences, Moscow
  - Russian National Research Medical University named after N.I. Pirogov, Moscow
  - Scientific Center for Children's Health of the Russian Academy of Medical Sciences, Moscow
  - Institute of the Human Brain named after N.P. Bekhtereva Russian Academy of Sciences, Saint Petersburg